CLINICAL TRIAL: NCT06341036
Title: Aetiology And Outcome Of Children With Thrombocytosis Admitted to Assiut University Children Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Mamdouh Safina Abid, Aetiology And Outcome Of children with Thrombocytosis admitted to Assiut University children hospital, Assiut University
Other Study IDs: Thrombocytosis in Children
Record Dates: First submitted 2024-02-19; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-01

CONDITIONS: Thrombocytosis in Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary Aim :to determine the etiology of thrombocytosis in children and frequency, outcome of thrombocytosis in Children.

DETAILED DESCRIPTION:
Thrombocytosis, also called thrombocythemia, is generally defined as a platelet count that is above the upper limit. The most commonly accepted cutoff value for normal is <450,000/μL. Platelet counts in the range of 450,000 to 700,000/μL are considered mild, between 700,000 and 900,000 /μL are considered moderate, between 900,000 and 1,000,000/μL are considered severe, and values above 1,000,000/μL are considered extreme thrombocytosis.The incidence of newly diagnosed primary thrombocytosis in children is about 1 per 10 million, about 60 times lower than adults.

The thrombocytosis is classified into primary thrombocytosis and secondary thrombocytosis. primary thrombocytosis classified into hereditary thrombocytosis which due to mutations in THPO,MPL,JAK2 and acquired primary thrombocytosis which classified into BCR-ABL1negative MPN as :Essential thrombocythemia(ET) , polycythemia vera(pv) ,primary myelofibrosis(PMF).and BCR-ABL1positive disorders but secondary thrombocytosis is due to :bacterial/viral infection,acute phase response ,chronic inflammation ,iron deficiency anemia , hemolytic anemia ,asplenia ,drugs :THPO analoga ,EPO.

Secondary thrombocytosis is commonly seen in children with a variety of clinical conditions. The most common cause of secondary thrombocytosis in children is respiratory infection .According to the World Health Organization guidelines, the persistent diagnosis of essential thrombocythemia requires a platelet count of ≥450,000/μL in patients with thrombocytosis, and it should be determined whether thrombocytosis is primary or secondary. The criteria of the World Health Organization are often used for diagnosis. .

In most cases, the symptoms are due to an underlying disorder and not the thrombocytosis itself. Extreme thrombocytosis may rarely result in thrombotic events such as acute myocardial infarction, mesenteric vein thrombosis, and pulmonary embolism.

The pathophysiology of thrombocytosis is according to each type:

Hereditary forms of primary thrombocytosis are caused by germline mutations within the genes encoding thrombopoietin (THPO), its receptor (MPL), and the receptor's effector kinase Januskinase2 (JAK2) .

Acquired primary thrombocytosis is marked by somatic mutations and occurs in several myeloid malignancies that are more commonly found in adults than in children. Therefore, most of the current knowledge on their pathogenesis and on their clinical management has been derived from studies in adults. Myeloid malignancies that may involve acquired primary thrombocytosis include myeloproliferative (MPNs) and myelodysplastic neoplasms (MDS), such as Philadelphia-positive chronic myeloid leukemia (CML), the Philadelphia-negative neoplasms ET, PV, and PMF, MPN/MDS with ring sideroblasts and thrombocytosis (RARS-T) or MDS with isolated del(5q) syndrome In secondary thrombocytosis , elevated platelet levels result from an extrinsic process, such as acute or chronic inflammation, which stimulates megakaryocytopoiesis . Thrombopoiesis is regulated by the interplay between thrombopoietin (THPO) and its receptor c-Mpl .In secondary thrombocytosis, interleukin-6 (Il-6) constitutes an additional key mediator .

ELIGIBILITY:
Inclusion Criteria:

all patients from age 1 month to 18 years old , who were admitted to Assiut University Children's Hospital with thrombocytosis

Exclusion Criteria:

1-Neonates ,Children with malignancy , 2_Children with polycythemia vera

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with Thrombocytosis
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-03-03 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Aetiology And Outcome Of children with Thrombocytosis admitted to Assiut University children hospital | Basalin
  Patient will be classified into two groups according to type primary and secondary. Each group will be compared :
  * demographically
  * clinically
  * on treatment and Outcome